CLINICAL TRIAL: NCT00556205
Title: Phase II, Randomized Trial of Bevacizumab With or Without Sunitinib in Sunitinib-Refractory Patients With Metastatic Renal Cell Carcinoma
Brief Title: Bevacizumab With or Without Sunitinib in Sunitinib-Refractory Renal Cell Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Toxicity of combination from other trials
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Dror Michaelson, MD, Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 07-202
Record Dates: First submitted 2007-11-07; First posted 2007-11-09 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Renal Cell Carcinoma
Keywords: mRCC; sunitinib; bevacizumab
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Bevacizumab monotherapy 10 mg/kg IV q2 weeks
  Interventions: Drug: Bevacizumab
- 2 (Active Comparator): Combination Sunitinib & Bevacizumab Bevacizumab 10 mg/kg IV q2 weeks Sunitinib 50 mg PO QD on 4/2 schedule
  Interventions: Drug: Sunitinib; Drug: Bevacizumab

INTERVENTIONS:
Drug: Sunitinib — Sunitinib orally once daily
  Other Names: sutent
  Arms: 2
Drug: Bevacizumab — Intravenously every 14 days
  Other Names: avastin

SUMMARY:
The purpose of this research study is to further define an effective strategy for people with renal cell carcinoma and to learn the safety and effectiveness of two different types of sunitinib-refractory treatments: Bevacizumab alone or a combination of sunitinib and bevacizumab. Sunitinib is an FDA approved drug and is currently one of the standard treatments for advanced renal cell carcinoma. However, some people who receive this treatment do not respond to treatment or they stop responding to treatment. Bevacizumab is an FDA approved drug used for the treatment of several cancers however, is not yet approved for use in renal cell carcinoma.

DETAILED DESCRIPTION:
* Participants will receive one of two treatment possibilities. Since no one knows which of the study options is best, participants will be "randomized" to one fo the three treatment groups.
* Group 1 will stop their current treatment with sunitinib and receive a dose of bevacizumab once every 2 weeks. Group 2 will receive the standard treatment of sunitinib with the addition of bevacizumab.
* All study participants will undergo the same study procedures. These study procedures will include the following at intervals specified in the protocol: medical history review; vital signs; physical exam; urine analysis; EKG and CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic renal cell carcinoma with clear cell histology
* Patients must be off sunitinib for 14 days prior to day 1 of treatment on protocol
* Evidence of unidimensionally measurable disease based on RECIST criteria, with at least 1 measurable lesion
* Radiographic evidence of disease progression defined by RECIST during or within 6 weeks of completion of sunitinib treatment
* Participants must have received at least 14 doses of sunitinib therapy
* Participants must enroll within 3 months of the last dose of sunitinib
* Males or females, age of 18 years or older
* ECOG Performance status 0-2
* Resolution of all acute toxic effects of prior therapy, radiotherapy or surgical procedures to NCI CTCAE version 3.0 grade 1 or less
* Laboratory values as defined in protocol
* 4 weeks or more must have elapsed from the time of major surgery and subjects must have recovered from the procedure prior to day 1 of randomization
* No anticipated need for major surgical procedure during the course of the study
* 2 weeks or more must have elapsed from the time of minor surgery and subjects must have recovered from the procedure prior to day 1 of randomization
* 4 weeks of more must have elapsed from the time of major radiotherapy prior to day 1 of randomization

Exclusion Criteria:

* Prior treatment with bevacizumab
* Unacceptable toxicity on prior sunitinib therapy at 37.5mg or lower
* Prior systemic therapy for RCC with > 2 regimens
* Systemic therapy other than sunitinib within 4 weeks of starting the study treatment
* Uncontrolled high blood pressure
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* History of abdominal fistula, gastrointestinal perforation or intraabdominal abscess within 3 months prior to day 0
* Any of the following within the 6 months prior to sudy drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, cerebrovascular accident or transient ischemic attack, symptomatic congestive heart failure, or ejection fraction < 30%
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range without medication
* History of or known brain metastases or spinal cord compression
* NCI CTCAE grade 2 or above hemorrhage within 4 weeks of starting study treatment
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Grade 3 or higher cardiac dysrhythmia or QT prolongation
* Concurrent use of proarrhythmic medications including terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide and flecainide
* Pregnancy or breastfeeding or inadequate contraception
* Significant thromboembolic event within 6 months
* Evidence of bleeding diathesis or coagulopathy
* Serious, non-healing wound, ulcer or bone fracture
* Proteinuria at screening
* Known hypersensitivity to any component of bevacizumab
* Psychiatric illness/social situation that would limit compliance with study requirements
* Previous or concurrent malignancy requiring active systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To determine the time to tumor progression (TTP) in this patient population treated with bevacizumab or combination of sunitinib and bevacizumab. | Until tumor progression

SECONDARY OUTCOMES:
To determine the overall response rate in this patient population. | Until tumor progression
To evaluate the safety and tolerability of these treatments in mRCC patients with disease progression on standard dose sunitinib. | Until tumor progression
To collect serum research samples for analysis of predictive biomarkers of response. | Two months

CONTACTS AND LOCATIONS:
Overall Officials: M. Dror Michaelson, MD, PhD, Principal Investigator — Massachusetts General Hosptial

IPD SHARING:
Plan to Share IPD: No
No data to share